CLINICAL TRIAL: NCT03308916
Title: Screening At-risk Populations for Hepatic Fibrosis With Non-invasive Markers
Acronym: SIPHON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maja Thiele (Other)
Collaborators: Horizon 2020 - European Commission (Other); Novo Nordisk A/S (Industry); University of Southern Denmark (Other); Esbjerg University Hospital of South-West Jutland (Unknown); Odense Municipality Alcohol Rehabilitation Unit (Unknown); Svendborg Municipality Alcohol Rehabilitation Unit (Unknown); University of Copenhagen (Other); University of Oslo (Other); Nordic Bioscience A/S (Industry); VLV Bio, Peviva AB (Unknown); Manatee APS (Unknown); Siemens Healthcare A/S (Industry); Steno Diabetes Center Copenhagen (Other); Biomedical Research Foundation, Academy of Athens (Other); European Molecular Biology Laboratory, EMBL, University of Heidelberg (Unknown)
Responsible Party: Sponsor-Investigator, Maja Thiele, Associate professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20170087
Record Dates: First submitted 2016-02-04; First posted 2017-10-13 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Liver Diseases, Alcoholic; Fibrosis
Keywords: elastography; screening; non-invasive markers; microbiome; gut-liver-axis; cost-benefit; fibroscan; aixplorer; ultrasound elastography; liver fibrosis; alcoholic liver disease; advanced fibrosis; enhanced liver fibrosis test; direct liver fibrosis markers; ELF; cytokeratin-18; neoepitopes; collagen; NAFLD; ALD; metabolomics; non-alcoholic fatty liver disease
MeSH Terms: conditions — Liver Diseases, Alcoholic; Fibrosis; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — Extracellular Polymeric Substance Matrix; Genome

STUDY DESIGN:
Intervention Model Description: Single intervention group selected for screening with a historical control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver stiffness measurement (Experimental): Transient elastography in fasting state
  Interventions: Diagnostic Test: transient elastography; Diagnostic Test: Enhanced liver fibrosis test; Diagnostic Test: Indirect serum markers of liver fibrosis; Diagnostic Test: Direct serum markers of liver fibrosis; Diagnostic Test: LiverTRAIL; Diagnostic Test: Cytokeratin 18; Diagnostic Test: Omics markers

INTERVENTIONS:
Diagnostic Test: transient elastography — Ultrasound elastography using shear-wave elastography to measure liver stiffness as a marker of liver fibrosis. Patients with transient elastography above 8.0 kPa selected for liver biopsy to detect advanced liver fibrosis
  Other Names: FibroScan; TE
Diagnostic Test: Enhanced liver fibrosis test — Patented, commercially available algorithm of hyaluronic acid (HA), N-terminal propeptide of collagen type 3 (P3NP) and tissue inhibitor of metalloproteinase 1 (TIMP-1)
  Other Names: ELF
Diagnostic Test: Indirect serum markers of liver fibrosis — Diagnostic markers using combination of routine liver biochemistry: age, AST, ALT, platelet count, cholesterol, GGT
  Other Names: Forns index; FIB-4; APRI; AST-ALT ratio; Age-platelet ratio
Diagnostic Test: Direct serum markers of liver fibrosis — Serum markers that reflect liver extracellular matrix turnover and -accumulation
  Other Names: Neoepitopes; Collagen products; Extracellular matrix
Diagnostic Test: LiverTRAIL — Software that contain 199 diagnostic algorithms, containing combinations of routine tests: age, AST, albumin, alkaline phosphatase, bilirubin, GGT, INR, platelet count, cholesterol and sodium, and specialist tests: transient elastography and direct serum markers of fibrosis.
Diagnostic Test: Cytokeratin 18 — Cytokeratin 18 from liver cell cytoskeleton; when cells undergo apoptosis, caspase-cleaved CK18 is released (M30), whereas full-length CK18 is realised during necrosis (M65)
  Other Names: CK18; M30; M65
Diagnostic Test: Omics markers — Markers combining signatures of liver fibrosis and hepatic inflammation from many 'omics technologies
  Other Names: Multi-omics markers; Lipidomics; Microbiomics; Genomics; Metagenomics; Metatranscriptomics; Transcriptomics; miRNA-omics; Metabolomics; Proteomics

SUMMARY:
Prospective screening study at Odense University Hospital to assess the effect of transient elastography and other serum and imaging markers of liver fibrosis to detect advanced fibrosis (Kleiner Fibrosis score F3-F4) in patients at risk of non-alcoholic fatty liver disease, alcoholic fatty liver disease, with a control group of participants recruited from the general population.

DETAILED DESCRIPTION:
This protocol describes a prospective screening study at Odense University Hospital, Department of Gastroenterology and Hepatology. The investigators will use liver stiffness measurements with transient elastography to screen 3000 participants from at-risk populations and 3500 participants from the general population for advanced liver fibrosis. At-risk is defined as either (A) a prior or current alcohol overuse (≥21 units/week for men and ≥14 units/week for women) for more than 5 years, or (B) presence of the metabolic syndrome with or without concomitant type 2 diabetes mellitus.

The study goal is to evaluate the aptitude of transient elastography as a screening tool for advanced liver fibrosis, based on analyses of benefit, harm, detection rate, technical applicability and prognostic potential. Secondary aims are to compare novel serum markers of liver fibrosis as potential screening tools against transient elastography: The Enhanced Liver Fibrosis test, neoepitope markers of extracellular matrix turnover, cytokeratin-18 based markers and indirect indices of fibrosis from algorithms combining routine liver blood test. Screened participants with elevated liver stiffness (≥8.0 kiloPascal; estimated 400 participants with alcoholic liver disease, 400 participants with non-alcoholic fatty liver disease and 280 participants from the general population) will be investigated with 2-dimensional shear-wave elastography and abdominal ultrasonography and a liver biopsy to confirm or reject presence of advanced fibrosis.

All participants with a positive screening elastography will be invited for repeated liver stiffness measurements and serum fibrosis markers after a minimum of one year from inclusion.

Participants at risk of alcoholic and non-alcoholic liver disease, independent of liver stiffness measurement at inclusion, will be invited for repeated liver stiffness measurements and serum fibrosis markers after a minimum of one year from inclusion. At-risk participants with elevated liver stiffness measurements at a follow-up visit (>6.0 kiloPascal) will be offered a liver biopsy, however no earlier than two years after the index biopsy.

All participants will be followed for 10 years to assess liver-related outcomes and all-course mortality.

ELIGIBILITY:
INCLUSION CRITERIA

Patients are eligible for screening if the following inclusion criteria are fulfilled:

* Age 30-75 years (except the general population, which should be aged 40-75)
* Informed consent to study investigations
* Ability to read and write Danish AND (only at-risk patients)
* Prior or current alcohol overuse, defined as an average intake of ≥24 grams/day (14 units/week) for women and ≥36 grams/day (21 units/week) for men, for at least 5 years; OR
* Presence of the metabolic syndrome defined by central obesity plus any two of the following four metabolic risk factors: (a) raised triglycerides, (b) reduced HDL cholesterol, (c) raised blood pressure and (d) raised fasting plasma glucose;[38] OR
* Type 2 diabetes mellitus defined by either fasting plasma glucose ≥7 mmol/L, HbA1c ≥48 mmol/mol, a random plasma glucose ≥11.1 mmol/L in the presence of classic diabetes or an oral glucose tolerance test with fasting plasma glucose ≥7.0 mmol/L and/or 2 hour plasma glucose ≥11.1 mmol/L.

EXCLUSION CRITERIA

We will exclude patients from screening in case of:

* Evidence of decompensated liver disease, defined by clinically obvious ascites, overt hepatic encephalopathy, jaundice or large esophageal varices with/without variceal bleeding.
* Known concurrent liver disease other than ALD and NAFLD.
* Cancer or other debilitating disease with an expected survival of less than 12 months.
* Inability to comply with the study protocol.

In screened patients with liver stiffness ≥8 kPa we will abstain from a liver biopsy in case of:

* Contraindications for a percutaneous liver biopsy
* Severe alcoholic hepatitis or other hepatic inflammation evidenced by transaminase elevation of more than three times the upper limit of normal.
* Hepatic congestion or bile duct dilation evidenced by ultrasound.
* Decrease of TE below 6.0 kPa from screening to time of planned liver biopsy.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2035-10-30 (Estimated)

PRIMARY OUTCOMES:
Biopsy-verified advanced fibrosis | 5 years
  Number of patients with biopsy-verified, advanced fibrosis (Kleiner fibrosis score ≥F3) detected by screening
Liver-related outcomes | 10 years
  Number of liver-related clinical outcomes during 10 years of follow up after the first screened patient, compared to a matched, historical control group (The Inter99 study and the Copenhagen and Odense alcohol rehabilitation cohorts). Liver-related outcomes are defined as liver-related death, liver transplant, progression to liver-related complications (ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, jaundice, bleeding from esophagastric varices, hepatocellular carcinoma) or MELD-Na score >15

SECONDARY OUTCOMES:
Liver related outcomes | 10 years
  Number of liver-related clinical outcomes during 10 years of follow up after the first screened patient, compared to a matched, historical control group (The Inter99 study and the Copenhagen and Odense alcohol rehabilitation cohorts). Liver-related outcomes are defined as liver-related death, liver transplant, progression to liver-related complications (ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, jaundice, bleeding from esophagastric varices, hepatocellular carcinoma) or MELD-Na score >15
Mortality | 10 years
  Overall number of deaths during 10 years of follow up after the first screened patient, compared to a matched, historical control group (The Inter99 study and the Copenhagen and Odense alcohol rehabilitation cohorts).

CONTACTS AND LOCATIONS:
Overall Officials: Maja Thiele, MD, PhD, Professor, Principal Investigator — Department of Gastroenterology and Hepatology, Odense University Hospital
Locations (1):
- Department of Gastroenterology and Hepatology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
OPEN - Odense Patient Exploratory data Network, managed by Odense University Hospital
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After publication of study results
Access Criteria: Accessible after contact to OPEN, who will pass on the request to primary investigator. No criteria.
URL: https://open.rsyd.dk/OpenProjects/da/openProject.jsp?openNo=475

REFERENCES:
- [Derived] Hansen CD, Hansen JK, Israelsen M, Andersen P, Pikkupeura LM, Lindvig KP, Stinson SE, Schnefeld HL, Tellerup J, Fogt M, Torp N, Kjaergaard M, Bech KT, Thorhauge KH, Johansen S, Spedtsberg I, Deluran E, Villesen IF, Detlefsen S, Hansen T, Krag A, Thiele M. Prevalence, severity and determinants of steatotic liver disease among individuals with metabolic and alcohol risk from the community. J Hepatol. 2025 Dec;83(6):1278-1291. doi: 10.1016/j.jhep.2025.06.020. Epub 2025 Jul 5. PMID 40618958
- [Derived] Kjaergaard M, Lindvig KP, Thorhauge KH, Andersen P, Hansen JK, Kastrup N, Jensen JM, Hansen CD, Johansen S, Israelsen M, Torp N, Trelle MB, Shan S, Detlefsen S, Antonsen S, Andersen JE, Graupera I, Gines P, Thiele M, Krag A. Using the ELF test, FIB-4 and NAFLD fibrosis score to screen the population for liver disease. J Hepatol. 2023 Aug;79(2):277-286. doi: 10.1016/j.jhep.2023.04.002. Epub 2023 Apr 21. PMID 37088311